CLINICAL TRIAL: NCT01478373
Title: DOVIGIST: Phase II Trial to Evaluate the Efficacy and Safety of Dovitinib (TKI258) in Patients With Gastrointestinal Stromal Tumors Refractory and/or Intolerant to Imatinib
Brief Title: Efficacy and Safety of Dovitinib in Patients With Gastrointestinal Stromal Tumors Refractory and/or Intolerant to Imatinib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTKI258AIC02; 2011-001725-24 (EudraCT Number)
Record Dates: First submitted 2011-11-16; First posted 2011-11-23 (Estimated); Results first posted 2015-08-10 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: GIST; Dovitinib
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dovitinib (TKI258) (Experimental): Patients will receive Dovitinib (TKI258) on an outpatient basis at the dose of 500 mg qd for 5 days followed by 2 days off, every week for cycle of 4 weeks (28d) until disease progression, unacceptable toxicity, or consent withdrawal.
  Interventions: Drug: Dovitinib (TKI258)

INTERVENTIONS:
Drug: Dovitinib (TKI258) — Oral Dovitinib (TKI258) as a gelatin capsule of 100 mg strength and dosed on a flat scale of 500 mg on a 5 days on /2 days off dosing schedule.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Dovitinib in patients with gastrointestinal stromal tumors refractory and/or intolerant to Imatinib

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed GIST of any anatomical location, which is 1) unresectable and/ or metastatic with documented disease progression while on therapy with imatinib or 2) surgically removed localized GIST, recurrent on adjuvant imatinib or recurrent within the first 3 months after discontinuation of adjuvant imatinib or 3) patients with unresectable and/or metastatic GIST intolerant to imatinib
* Positive immunohistochemical staining for c-KIT (CD117); or negative staining for KIT, but with either positive staining for DOG1 or an identified mutation of KIT or PDGFRA gene
* Documented disease progression according to RECIST (version 1.1) on prior therapy with imatinib at a dose of at least 400mg/day or patients with unresectable and/or metastatic GIST who are intolerant to imatinib
* At least one measurable GIST lesion according to RECIST (version 1.1).
* Adequate bone marrow, liver and renal function

Exclusion Criteria:

* Patients who have received any other tyrosine-kinase inhibitor but imatinib for GIST
* Patients who received cytotoxic drugs ≤ 4 weeks prior to starting Dovitinib (TKI258)
* Patients who are treated or planned to be treated concomitantly with other cytotoxic or antineoplastic treatments, such as chemotherapy, immunotherapy, biological response modifiers, or radiotherapy
* Patients with another primary malignancy within 3 years prior to starting the study drug
* Patients who have undergone major surgery (e.g. intra-thoracic, intra-abdominal or intra-pelvic) ≤ 4 weeks prior to starting Dovitinib (TKI258) or who have not recovered from the adverse effects of such therapy
* Patients with a history of pulmonary embolism (PE), or untreated deep venous thrombosis (DVT) within the past 6 months
* Patients with impaired cardiac function or clinically significant cardiac diseases
* Patients with impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of Dovitinib
* Patients with prior complete gastrectomy
* Patients with brain metastasis or history of brain metastasis
* Patients who are currently receiving anticoagulation treatment with therapeutic doses of warfarin or equivalent anticoagulant
* Pregnant or breast-feeding women

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2012-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Study Director, Study Director — Novartis Pharmaceuticals
Locations (15):
- Novartis Investigative Site, HUS, Finland
- France (5):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Villejuif
- Novartis Investigative Site, Essen, Germany
- Italy (4):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Candiolo, TO
  - Novartis Investigative Site, Torino, TO
- Spain (4):
  - Novartis Investigative Site, Palma de Mallorca, Balearic Islands
  - Novartis Investigative Site, Barcelona, Barcelona
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 39 Patients enrolled. One patient had a protocol deviation which excluded him from the Full Analysis Set.
Groups:
- Dovitinib: Patients received Dovitinib (TKI258) on an outpatient basis at the dose of 500 mg qd for 5 days followed by 2 days off, every week for cycle of 4 weeks (28d) until disease progression, unacceptable toxicity, or consent withdrawal.
Period: Treatment Phase
Arm/Group | Dovitinib
Started | 39
Completed | 38
Not Completed | 1
Not completed — Protocol Violation | 1
Period: Survival Phase
Arm/Group | Dovitinib
Started | 38
Completed | 0
Not Completed | 38
Not completed — Adverse Event | 8
Not completed — Protocol Violation | 1
Not completed — crossover to another study | 2
Not completed — Progressive Disease | 27

BASELINE CHARACTERISTICS:
Population: Full Analysis Set - All subjects with histologically confirmed diagnosis of GIST who received at least one dose of study drug.
Arm/Group | Dovitinib
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.2 (10.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 22

OUTCOME MEASURES:

1. Primary Outcome: Antitumor Activity of Dovitinib in Terms of Disease Control Rate (DCR): Complete Response+Partial Response +Stable Disease
Description: DCR is defined as the proportion of patients with a best overall response of Complete Responses (CR), Partial Response (PR) and Stable Disease (SD) at 12 weeks according to RECIST (version 1.1). Complete Response (CR): Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm 1;Partial Response (PR): At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters. Progressive Disease (PD): At least a 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm2. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for PD.
Time Frame: 12 Weeks
Population: Full Analysis Set: all subjects with histologically confirmed diagnosis of GIST who received at least one dose of study drug.
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Dovitinib
Number analyzed (Participants) | 38
Percentage of Participants | 52.6 [38.2 to 66.7]

2. Secondary Outcome: Progression-free Survival (PFS) of Patients Treated With Dovitinib
Description: The PFS duration: time from entry into the study to the date of the first documented progression (assessed using conventional RECIST (version 1.1) or death due to any cause. Progression is defined using Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 9 months
Population: as for outcome 1
Measure: Median (90% Confidence Interval); unit: Days
Arm/Group | Dovitinib
Number analyzed (Participants) | 38
Days | 141 [86.0 to 225.0]

3. Secondary Outcome: Time to Treatment Failure (TTF)of Patients Treated With Dovitinib
Description: TTF: the date of entry into the study to the earliest date of the first objective tumor progression, date of death due to any cause, or date of discontinuation due to reasons other than 'Protocol deviation' or 'Administrative problems'.
Time Frame: 9 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Dovitinib
Number analyzed (Participants) | 38
Days | 122.0 [81.0 to 223.0]

4. Secondary Outcome: Duration of Response or Stable Disease (SD)
Description: Duration of response or SD: time from date of entry into study to earliest date of first objective tumor progression or death. DCR is defined as proportion of patients with best overall response of CR, PR and SD at 12 weeks according to RECIST (version 1.1). CR: Disappearance of all non-nodal target lesions. Any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm 1; PR: At least a 30% decrease in sum of diameter of all target lesions, taking as reference the baseline sum of diameters. PD: At least a 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm2. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for PD.
Time Frame: 9 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Dovitinib
Number analyzed (Participants) | 38
Days | 193.2 (117.78)

5. Secondary Outcome: Time to Tumor Progression (TTP)of Patients Treated With Dovitinib
Description: TTP: time from the date of entry into the study to first documentation of tumor progression or death due to the underlying cancer. Progression is defined using Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 9 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Dovitinib
Number analyzed (Participants) | 38
Days | 141.0 [85.0 to 229.0]

6. Secondary Outcome: Overall Response Rate (ORR) of Patients Treated With Dovitinib
Description: Outcome Measure Description: ORR: proportion of patients whose best overall response is either complete response (CR) or partial response (PR) according to RECIST (version 1.1). Complete Response (CR): Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm 1;Partial Response (PR): At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters. Progressive Disease (PD): At least a 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm2. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for PD.
Time Frame: Baseline, 12 weeks
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Dovitinib
Number analyzed (Participants) | 38
Percentage of Participants | 2.6 [0.1 to 11.9]

7. Secondary Outcome: Overall Survival (OS) of Patients Treated With Dovitinib
Description: Outcome Measure Description: OS: time from the date of entry into the study to the date of death due to any cause. A patient who has not died by the date of the analysis cut-off would have the OS censored at the time of the last contact before the cut-off date.
Time Frame: 21 months (9 months of estimated treatment plus 12 months of survival follow up)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dovitinib
Number analyzed (Participants) | 38
Months | NA [NA to NA] — The median survival had not been reached

8. Secondary Outcome: DCR (CR+PR+SD) at the End of Treatment
Description: DCR is defined as the proportion of patients with a best overall response of CR, PR and SD at the end of dovitinib treatment according to RECIST (version 1.1). Complete Response (CR): Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm 1;Partial Response (PR): At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters. Progressive Disease (PD): At least a 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm2. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for PD.
Time Frame: Up to 9 months of estimated treatment
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Dovitinib
Number analyzed (Participants) | 38
Percentage of Participants | 52.6 [38.2 to 66.7]

ADVERSE EVENTS:
Arm/Group | Dovitinib
Serious Adverse Events (participants affected / at risk) | 16/39
Other Adverse Events (participants affected / at risk) | 36/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dovitinib (N=39)
Anaemia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Asthenia (General disorders) | 1
Fatigue (General disorders) | 4
General physical health deterioration (General disorders) | 1
Inflammation (General disorders) | 1
Localised oedema (General disorders) | 1
Mucosal dryness (General disorders) | 1
Oedema peripheral (General disorders) | 1
Systemic inflammatory response syndrome (General disorders) | 1
Cholestasis (Hepatobiliary disorders) | 1
H1N1 influenza (Infections and infestations) | 1
Tracheobronchitis (Infections and infestations) | 1
Red blood cell count decreased (Investigations) | 1
Weight decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Mania (Psychiatric disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1
Aortic thrombosis (Vascular disorders) | 1
Phlebitis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dovitinib (N=39)
Anaemia (Blood and lymphatic system disorders) | 6
Neutropenia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Tinnitus (Ear and labyrinth disorders) | 2
Vertigo (Ear and labyrinth disorders) | 3
Dry eye (Eye disorders) | 2
Keratitis (Eye disorders) | 3
Lacrimation increased (Eye disorders) | 6
Ocular hyperaemia (Eye disorders) | 2
Periorbital oedema (Eye disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 11
Abdominal pain upper (Gastrointestinal disorders) | 8
Constipation (Gastrointestinal disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 28
Dry mouth (Gastrointestinal disorders) | 6
Dyspepsia (Gastrointestinal disorders) | 3
Gastric disorder (Gastrointestinal disorders) | 3
Haemorrhoids (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 17
Stomatitis (Gastrointestinal disorders) | 2
Toothache (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 21
Asthenia (General disorders) | 15
Chest pain (General disorders) | 4
Fatigue (General disorders) | 14
Malaise (General disorders) | 3
Mucosal inflammation (General disorders) | 4
Oedema peripheral (General disorders) | 3
Pyrexia (General disorders) | 7
Hepatocellular injury (Hepatobiliary disorders) | 2
Nasopharyngitis (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Alanine aminotransferase increased (Investigations) | 10
Aspartate aminotransferase increased (Investigations) | 11
Blood alkaline phosphatase increased (Investigations) | 13
Blood bilirubin increased (Investigations) | 4
Blood calcium decreased (Investigations) | 2
Blood lactate dehydrogenase increased (Investigations) | 3
Blood triglycerides increased (Investigations) | 2
C-reactive protein increased (Investigations) | 2
Gamma-glutamyltransferase increased (Investigations) | 14
Lipase increased (Investigations) | 4
Protein total decreased (Investigations) | 2
Weight decreased (Investigations) | 12
Decreased appetite (Metabolism and nutrition disorders) | 15
Dyslipidaemia (Metabolism and nutrition disorders) | 3
Hypercholesterolaemia (Metabolism and nutrition disorders) | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 13
Hypoalbuminaemia (Metabolism and nutrition disorders) | 7
Hypocalcaemia (Metabolism and nutrition disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7
Dysaesthesia (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 6
Headache (Nervous system disorders) | 8
Neuropathy peripheral (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 6
Sciatica (Nervous system disorders) | 4
Anxiety (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 4
Sleep disorder (Psychiatric disorders) | 2
Pollakiuria (Renal and urinary disorders) | 4
Proteinuria (Renal and urinary disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 8
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 6
Deep vein thrombosis (Vascular disorders) | 2
Hypertension (Vascular disorders) | 13
Hypotension (Vascular disorders) | 2
Tachicardia (Cardiac disorders) | 2
Ascites (Gastrointestinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.